CLINICAL TRIAL: NCT05245773
Title: MORE-PC: A 30-day Automated SMS Program to Support Post-discharge Transitions of Care
Acronym: MORE-PC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: UnitedHealth Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 849348
Record Dates: First submitted 2022-02-08; First posted 2022-02-18 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Care Transitions
Keywords: Post-Discharge; Primary Care; Automated Hovering

STUDY DESIGN:
Intervention Model Description: Pragmatic randomized controlled trial with intervention and control arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30-day automated hovering + usual care (Experimental): The intervention arm will get the usual post-discharge call from their practice, typically within 2 business days of discharge. In addition, they will be enrolled in the 30-day automated texting program, wherein they will receive check-in messages on a tapering schedule; they will be free to opt out at any time. They can also message into the platform at any time. Any needs identified through the platform will be escalated to their primary care practice, and they will receive a follow-up phone call from practice staff to address their needs.
  Interventions: Other: Automated SMS program to support post-discharge transitions of care
- Usual care (No Intervention): The control arm will continue to receive the usual post-discharge call from their practice, typically within 2 business days of discharge.

INTERVENTIONS:
Other: Automated SMS program to support post-discharge transitions of care — The intervention will consist of automated text messages on a tapering schedule over the course of 30 days post-discharge, with responses escalated back to the practice care management team. After initial enrollment messages, patients will receive check-in messages on a tapering schedule over the course of 30 days. For the first week they will receive 3 total messages; the second week they will receive a total of 2 messages. For the last 2 weeks they will receive weekly messages. If a patient need is identified, the request will be escalated to the practice (triaged by the care management RN) for a follow up phone call. Patients will be able to reach out at any time by sending a message to the same number, and they will be entered into the same pathway. For any escalated need, patients will receive a follow up phone call from the practice staff.
  Other Names: MORE-PC
  Arms: 30-day automated hovering + usual care

SUMMARY:
This study will evaluate a 30-day post-discharge intervention using an automated SMS platform to monitor patients and facilitate communication with their primary care practice. The population will be patients who receive care from participating practices and are discharged from an inpatient stay. In addition to the usual phone call from their practice, patients will be randomized to enrollment in the program, wherein they will receive automated SMS messages on a tapering schedule over 30 days.

DETAILED DESCRIPTION:
Background:

Current models of post-discharge care management are time and labor intensive, limited in scope, and inconvenient from the patient perspective, particularly when they have a need arise. Automation can significantly scale up patient touches while reserving staff time for concrete patient needs. Text messaging has been shown to enhance patient engagement (as compared to calls) in many settings, possibly due to greater convenience and the potential for asynchronous interaction. We believe using automated text messaging messaging as the foundation of a post-discharge, primary care based care management program can increase patient engagement, allow for earlier and more frequent identification of needs, and improve post-discharge outcomes.

Objective:

To evaluate the impact of a 30-day post-discharge intervention using an automated SMS platform in addition to usual care as compared to usual care alone in a multi-clinic, pragmatic randomized controlled trial on acute care utilization, post-discharge follow-up appointment scheduling and show-rates, overall patient engagement, and overall patient-clinic encounters.

Description of Intervention:

The intervention will consist of automated text messages on a tapering schedule over the course of 30 days post-discharge, with responses escalated back to the practice care management team. After enrollment, patients will receive an initial message asking them if they have a follow up appointment within the next 2 weeks. If they respond no, the practice will be notified to reach out and help them schedule an appointment.

Beginning the day after this introductory message, patients will receive check-in messages on a tapering schedule over the course of 30 days. For the first week they will receive 3 total messages (Monday, Wednesday and Friday); the second week they will receive a total of 2 messages (Tuesday and Thursday). For the last 2 weeks they will receive weekly messages (on Tuesdays). If a patient need is identified, the request will be escalated to the practice (triaged by the care management RN) for a follow up phone call. Patients will be able to reach out at any time throughout the 30 days by sending a message to the same number, and they will be entered into the same pathway. For any escalated need, patients will receive a follow up phone call within 1 business day. Patients who do not respond to 3 consecutive messages will receive an additional check in message ensuring that they still want to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

* The study subjects will be medium to high risk (UPHS risk score 4 and above; an internally developed and validated score assessing a patient's risk for readmission) adult (age ≥ 18) patients of the Penn Primary Care Practices who are discharged home from acute inpatient care in the broad Philadelphia region as identified in HealthShare Exchange (HSX) reports

Exclusion Criteria:

* This study will exclude discharges who do not meet criteria for transitional care management. These criteria include discharges after 1) planned chemotherapy admissions; 2) certain scheduled surgeries, including spinal surgery, joint replacements, gastric bypass, transurethral resection of the prostate, gynecologic surgeries, and transplants; 3) obstetrics admissions.
* We will exclude patients from re-enrollment during the study period (once they have been enrolled once, they will not be enrolled again). We will also exclude patients being discharged to home hospice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5000 (Actual)
Dates: Start 2022-03-29 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Post-discharge acute care utilization | 30 days post-discharge
  A composite, binary measure indicating whether a patient visited the ED or was readmitted to inpatient care after discharge from the hospital.

SECONDARY OUTCOMES:
Post-discharge days in the hospital | 30 days post-discharge
  A continuous measure of total days spent in the hospital (in the ED or as an inpatient) after hospital discharge
Post-discharge acute care utilization | 7 and 60 days post-discharge
  A composite, binary measure indicating whether a patient visited the ED or was readmitted to inpatient care after discharge from the hospital.
Post-discharge ED visit | 7, 30, and 60 days post-discharge
  A binary measure indicating whether a patient visited the ED after hospital discharge
Readmission | 7, 30, and 60 days post-discharge
  A binary measure indicating whether a patient was readmitted after hospital discharge
Time from discharge to first acute care visit | 30 days post-discharge
  A continuous measure of the time from discharge to either first ED visit or readmission
Post-discharge follow up visit | 14 days post-discharge
  A binary measure indicating scheduling and completion of a follow up visit with the primary care practice
Number of patient-practice interactions | 30 days post-discharge
  A continuous measure of non-visit interactions between the patient and practice (which will include a) telephone encounters [which are the end point of any needs identified through the automated messaging program] and b) EMR portal messages)

CONTACTS AND LOCATIONS:
Overall Officials: Anna Morgan, MD, MSHP, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Bressman E, Long JA, Burke RE, Ahn A, Honig K, Zee J, McGlaughlin N, Balachandran M, Asch DA, Morgan AU. Automated Text Message-Based Program and Use of Acute Health Care Resources After Hospital Discharge: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e243701. doi: 10.1001/jamanetworkopen.2024.3701. PMID 38564221